CLINICAL TRIAL: NCT04211506
Title: Comparison Across Multiple Types of Sleep Deprivation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Civil Aerospace Medical Institute (U.S. Federal Agency)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: GEN10025
Record Dates: First submitted 2019-12-05; First posted 2019-12-26 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Sleep Deprivation; Sleep Restriction
Keywords: Neurobehavioral performance; Genetic
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Intervention Model Description: Each participant will undergo one of four separate arms manipulating levels and timing of sleep in a controlled laboratory setting.
Who Masked: Participant
Masking Description: Participants may not know to which study arm they are assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sleep Arm 1 (Experimental): This will be the first of four arms of controlled sleep manipulation.
  Interventions: Behavioral: Controlled sleep
- Sleep Arm 2 (Experimental): This will be the second of four arms of controlled sleep manipulation.
  Interventions: Behavioral: Controlled sleep
- Sleep Arm 3 (Experimental): This will be the third of four arms of controlled sleep manipulation.
  Interventions: Behavioral: Controlled sleep
- Sleep Arm 4 (Experimental): This will be the fourth of four arms of controlled sleep manipulation.
  Interventions: Behavioral: Controlled sleep

INTERVENTIONS:
Behavioral: Controlled sleep — Duration and timing of sleep will be assigned and monitored in a controlled laboratory environment with controlled lighting and meals.

SUMMARY:
This study is designed to assess neurobehavioral performance, as well as genetic and other physiological changes associated with variations in timing and quantity of sleep.

DETAILED DESCRIPTION:
During a 1.5 week inpatient laboratory protocol, subjects will undergo one of four parallel sleep conditions. Subjects will be randomly assigned to each condition group. During their time in the laboratory, biological samples (e.g., blood) will be collected for genetic and other analyses, and sleep quantity and quality will be monitored. Additionally responses on neurobehavioral tests and surveys will be monitored for differences among the groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* BMI 18.5-29.9, with consideration of BMIs 30-34.9.

Exclusion Criteria:

* Medication use, with potential consideration for contraceptives.
* Color blindness
* Recent nightwork, shiftwork, or travel across greater than two time zones
* Pregnant or within 6 months post-partum

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Gene expression changes associated with different sleep patterns. | Samples for gene expression will be collected at frequent intervals over 10 days in a sleep laboratory. Subjects will be in a time-free environment, and not told sampling frequency.
  Levels of expression of all genes may be compared across time and among study arms with different sleep patterns using RNA-Seq and differential expression analysis with generalized linear models. Patterns may be sought with and potential relevance to sleep, circadian rhythms, and/or neurobehavioral performance.

SECONDARY OUTCOMES:
Neurobehavioral performance changes associated with different sleep patterns. | Neurobehavioral assays may be conducted at frequent intervals over 10 days in a sleep laboratory. Subjects will be in a time-free environment, and not told assay frequency.
  Neurobehavioral performance may be compared across time and among study arms with different sleep patterns. Specifically, differences will be examined in subjective and objective neurobehavioral assays (Karolinska sleepiness scale, Performance effort and evaluation rating scale, Digit symbol substitution test, Stroop performance, Raven matrix task, Comparative visual search, Face-name task, Psychomotor vigilance test, Visual analog scale, Track test, and the Balloon analog risk task). Patterns may be sought with relevance to sleep, circadian rhythms, and/or other outcome measures.
DNA genetic variants associated with sleep and/or neurobehavioral performance. | Approximately two oral samples may be taken for DNA analyses during the 10 days in a sleep laboratory.
  Analysis of genetic variants may be used to assess inherited genetic differences among subjects and potential relevance to sleep, circadian rhythms, and/or neurobehavioral performance.

OTHER OUTCOMES:
Microbiome metrics associated with sleep and/or neurobehavioral performance. | Approximately three fecal samples will be collected over the 10 days in a sleep laboratory for potential future microbiome analyses.
  Fecal samples will be collected and may be analyzed in the future for microbiome differences among subjects, over time, and/or with respect to study conditions and metrics (e.g., differences in microbiome associated with sleep and/or neurobehavioral performance).
Metabolite and protein metrics associated with sleep and/or neurobehavioral performance. | A series of blood samples will be collected over the 10 days in a sleep laboratory for potential future analyses.
  Blood samples will be collected and may be analysed in the future for metabolite, protein, or other molecular differences among subjects, over time, and/or with respect to study conditions and metrics (e.g., differences associated with sleep and/or neurobehavioral performance).
Additional urine and saliva | Saliva and urine samples will be collected frequently during wake over the 10 days in a sleep laboratory for potential future analyses
  Urine and saliva samples will be collected and may be analyzed in the future for metabolite, protein, or other genetic differences among subjects, over time, and/or with respect to study conditions and metrics
Additional physiological metrics. | Frequent data collection will be made prior to and during the 10 days in a sleep laboratory, including approximately 3 nights of polysomnography.
  Actigraphy, polysomnography, screening data and log/diary information will be collected and may be analysed in the future for comparison with other outcome measures, and particularly associations with sleep, circadian rhythms, and/or neurobehavioral performance.

CONTACTS AND LOCATIONS:
Overall Officials: Hilary Uyhelji, PhD, Principal Investigator — FAA Civil Aerospace Medical Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - FAA Civil Aerospace Medical Institute, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: Yes
Raw genetic data that form the basis of a manuscript are expected to be made available after publication in accordance with federal and IRB policy and restrictions.
Supporting Information: ICF
Time Frame: Release of genetic data forming the basis of a manuscript are expected to be made available after publication. Release will be consistent with Institutional Review Board, journal, and federal requirements.
Access Criteria: Access may be controlled, e.g., in accordance with the National Institutes of Health database of Genotypes and Phenotypes (dbGAP) controlled access policy.

REFERENCES:
- [Derived] Uyhelji HA, Nicholson SJ, Nesthus TE, Beckel JL, Klerman EB, Czeisler CA, Yuan RK, Arrona-Palacios A, Song P, Ronda JM, Goodson MS. Exploratory development of biomarkers for neurobehavioral performance impairment during sleep loss: comparison across multiple types of sleep deprivation. BMC Genomics. 2025 Nov 14;26(1):1043. doi: 10.1186/s12864-025-12193-6. PMID 41239200

DOCUMENTS (1):
  • Informed Consent Form (2023-01-12): https://cdn.clinicaltrials.gov/large-docs/06/NCT04211506/ICF_000.pdf